CLINICAL TRIAL: NCT02366624
Title: Effect of Gastric Bypass, Sleeve Gastrectomy and Duodenal-jejunal Bypass on Bile Acid Homeostasis
Brief Title: Effect of Bariatric Surgery on Bile Acid Homeostasis
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Sponsor
Other Study IDs: 11-126
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — * Blood samples (serum and plasma).
  * Stool samples.
  * Liver samples.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the effect of bariatric surgery in bile acid homeostasis and its interrelationship with the metabolic changes induced by the surgery.

This study contemplates the following hypothesis:

* Bariatric Surgery induce a new study state in bile acid homeostasis with higher bile acid synthesis in association with increased bile acid content.
* The major effects of bariatric surgery on bile acid synthesis and is observed one month after surgery with a progressively decline during the first year of follow-up.
* Gastric bypass increases serum bile acid content, postprandial plasma bile acid response and fecal bile acid excretion.
* Serum bile acids changes induced by gastric bypass are positively correlated with changes in gastric inhibitory polypeptide (GIP) levels and postprandial concentration of insulin and glucagon like peptide-1 (GLP-1) and inversely correlated with thyrotropic hormone (TSH) and postprandial concentration of glucose.
* Changes in postprandial plasma bile acid response induced by gastric bypass positively correlates with changes in postprandial concentration of insulin, GLP-1 and peptide YY (PYY) and inversely correlates postprandial response of ghrelin and glucose.

DETAILED DESCRIPTION:
The proposed study will be conducted in adult subjects that will undergo to gastric bypass,sleeve gastrectomy or endoscopic duodenal-jejunal bypass.

as treatment for their obesity. As a first approach (Protocol A) in each of these groups the investigators will determine 7α-hydroxy-4-cholestene -3-one (C4) levels, a marker of bile acid synthesis, and fibroblast growth factor 19 (FGF19), inhibitor of the expression of Cholesterol 7- hydroxylase (CYP7A1), prior to surgery and then at months 1, 3, 6 and 12 of postoperative follow-up. The same measurements will be performed to a group of patients under medical treatment when they achieve 10-kg diet-induced weight loss, which is equivalent to one-month of surgically induced weight loss. Preliminary studies suggest that gastric bypass induces a greater weight loss and improvement of associated disease compared with sleeve gastrectomy and endoscopic duodenal-jejunal bypass. Therefore, we expect a deeper change in bile acid homeostasis after gastric bypass, than after the other procedures. For this reason, in patients with gastric bypass the investigators will determine fecal excretion, synthesis, bile acid pool composition, and postprandial plasma response (Protocol B). These variables will be measured prior to surgery and one month after the procedure and also to the group of patients under medical treatment after a 10-kg diet-induced weight loss.

The expression of diverse enzymes, nuclear receptors, transcription factors, transporters as well as cell surface receptors will be quantified at messenger ribonucleic acid (mRNA) and protein level in liver biopsy samples obtained from patients at the time of gastric bypass or sleeve gastrectomy (Protocol C). Those parameters will be reevaluated in liver samples obtained from the same subjects within the first 12 months of the postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female, 18 to 50 years old.
* Body mass index(BMI)≥35 and <40 with comorbidities or BMI ≥40 and <45 with or without comorbidities.
* HbA1c<8%.
* Subjects willing to comply with study requirements.

Exclusion Criteria:

* Previous cholecystectomy or gallbladder stones at baseline visit.
* Previous bariatric surgery, small bowel or colon resection.
* Use of drugs:cholestyramine,colesevelam,colestilan, colestimide, colestipol,insulin,exenatide, thiazolidinedione or dipeptidyl peptidase IV(DPPIV)inhibitors, selective serotonin re uptake inhibitor antidepressants.
* Pregnancy or intent to become pregnant.
* Cardiac, renal or liver failure.
* Cancer,infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese patients that have undergone bariatric surgery or medical treatment to lose weight.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Analysis of hormones and bile acids in patients that have undergone bariatric surgery | One year

CONTACTS AND LOCATIONS:
Overall Officials: Alex G. Escalona, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile